CLINICAL TRIAL: NCT02739464
Title: Randomized, Controlled, Multicenter Study of the Effect of In-Patient Exercise Training on Length of Hospitalization, Mental Health, and Physical Performance in Burned Patients
Brief Title: Effect of In-Patient Exercise Training on Length of Hospitalization in Burned Patients
Acronym: MP-10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: United States Army Institute of Surgical Research (U.S. Federal Agency); University of Texas Southwestern Medical Center (Other); California State University, Sacramento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHC; IRB #14-0432
Record Dates: First submitted 2015-03-12; First posted 2016-04-15 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Muscle Weakness; Late Effect of Burn; Muscle; Fatigue, Heart; Burn Rehabilitation
Keywords: Burn; Exercise; Ergometer; MP-10
MeSH Terms: conditions — Muscle Weakness; Fatigue; Burns; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + SOC PT/OT (Experimental): SOC treatment plus a personalized, structured, and quantifiable exercise program (MP10) carried out soon after admission until hospital discharge (including during the BICU stay and time on ventilation.
  Interventions: Other: Exercise + SOC PT/OT
- SOC PT/OT (Active Comparator): Only SOC for treating in-patient burn subjects
  Interventions: Other: SOC PT/OT

INTERVENTIONS:
Other: Exercise + SOC PT/OT
  Arms: Exercise + SOC PT/OT
Other: SOC PT/OT
  Arms: SOC PT/OT

SUMMARY:
This study will measure efficacy of early in-patient exercise as an adjunct to current Standard of Care (SOC) for 96 patients in a multi-centre trial. The secondary purpose is to assess the efficacy of a personalized, structured, and quantifiable exercise program (MP10) carried out soon after admission until hospital discharge (including during the BICU stay and time on ventilation).

DETAILED DESCRIPTION:
After severe burns (≥ 30% total body surface area [TBSA] burns, patients enter a persistent and extensive hypermetabolic and catabolic state. Unfortunately, burn-induced muscle catabolism is exacerbated by the prolonged bed rest and inactivity that accompanies hospitalization, leading to further loss of muscle mass and extreme weakness. The persistence of weakness, fatigue, and muscle catabolism from prolonged bed rest and inactivity during the acute care stage ultimately delays rehabilitation and return to normal physical activities. Studies conducted in non-burn patients have shown that, aside from decreasing muscle mass, prolonged bed rest has a host of other negative physiological consequences.

The primary purpose of this randomized, controlled, multicenter study is being conducted to determine the efficacy of early in-patient exercise, when used as an adjunct to standard of care (SOC), in improving recovery of adults from burns. The secondary purpose is to assess the efficacy of a personalized, structured, and quantifiable exercise program (hereafter referred to as MP10) carried out soon after admission until hospital discharge (including during the BICU stay and time on ventilation). This objective will be met through a multicenter trial in children and adults (7 - 60 years) with ≥30% TBSA burns. Outcome variables will include BICU days, ventilator days, hospital days, peak treadmill time, and lean body mass and psychosocial function (See Section 8 for details).

Methods: Ninety-six subjects will be recruited from four sites (24 subjects each) for this study and all genders and ethnicities will be invited. All subject will have TBSA > 30% and be ages 7-60 years of age. The first objective of this multicenter study will be to characterize the SOC related to physical/occupational therapy of inpatients at four U.S. burn centers, through 25 question surveys. The second portion of the project will involve exercise research. The objective is to assess the efficacy of MP10, in conjunction with existing SOC, in reducing debilitation among discharged burn patients. This will be initiated following surgeon's prescription, roughly 3-5 days following the first surgery after admission.

Ergonomic exercise training for the in-patient subjects will be conducted using Leg and Arm Ergometer equipment, and the training period will be daily for 10 minutes. The duration will be the duration the patient is held in the Burn Intensive Care Unit (BICU). Testing will include the following: Lean mass (assessed via dual energy x-ray absorptiometry (DEXA), Cardiopulmonary and muscle endurance test (peak VO2 on treadmill test), and weekly 6 minute walk test.

Data Analysis: A repeated measure ANOVA will be calculated using lean body mass and peak VO2 as dependent variables with the independent variables of TBA%, duration of hospital stay (and days of ergonomic exercise), ventilator days, and demographics. The purpose of this study is to measure efficacy of exercise training while in BICU for thermal injury patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥7 to 60 years of age
2. >30% TBSA burned, as estimated by the physician in charge
3. No evidence of organ failure

Exclusion Criteria:

1. Active Tuberculosis- based on clinical symptoms and/or abnormal chest x-ray in the upper lobe.
2. Electrical burns
3. Mental retardation or autism or any other mental disorder that makes it impossible to participate in an exercise program
4. Pregnancy

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
change in lean muscle mass | It is the change from baseline until discharge. Baseline is the time in the ICU, approximately 1-3 months post burn. Discharge is within 3 weeks of the discharge date from the burn ICU. Study duration is at most 5 months depending on the patients burn.
  Kilograms

SECONDARY OUTCOMES:
change in VO2 max | It is the change from baseline until discharge. Baseline is the time in the ICU, approximately 1-3 months post burn. Discharge is within 3 weeks of the discharge date from the burn ICU. Study duration is at most 5 months depending on the patients burn.]
  The maximal amount of oxygen per kilogram of body mass per minute(ml/kg/min) in a cardiopulmonary exercise test.
change in distance walked over 6 minutes | It is the change from baseline until discharge. Baseline is the time in the ICU, approximately 1-3 months post burn. Discharge is within 3 weeks of the discharge date from the burn ICU. Study duration is at most 5 months depending on the patients burn.
  6 min walk test measures distance will be recorded in feet.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Suman, Principal Investigator — University of Texas Medical Branch/Shriners Hospital for Children
Locations (4):
- United States (4):
  - University of California-Davis/Shriners Hospitals for Children-Sacramento, Davis, California
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch/Shriners Hospitals for Children-Galveston (lead site), Galveston, Texas
  - United States Army Institute of Surgical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
ONLY de-identified data will be deposited with main site (UTMB). Subsequently, if data is shared among all sites, it will be always in de-identified manner and stripped of all information that could identify the participant.
Time Frame: Data will become available once study is completed and 7 years after that date, according to the IRB standards.
Access Criteria: Once study personnel has completed CITI training and add to the study, will they have access to the data.

REFERENCES:
- [Background] Bloomfield SA. Changes in musculoskeletal structure and function with prolonged bed rest. Med Sci Sports Exerc. 1997 Feb;29(2):197-206. doi: 10.1097/00005768-199702000-00006. PMID 9044223
- [Background] Bartone PT. Test-retest reliability of the dispositional resilience scale-15, a brief hardiness scale. Psychol Rep. 2007 Dec;101(3 Pt 1):943-4. doi: 10.2466/pr0.101.3.943-944. PMID 18232452
- [Background] Kildal M, Andersson G, Fugl-Meyer AR, Lannerstam K, Gerdin B. Development of a brief version of the Burn Specific Health Scale (BSHS-B). J Trauma. 2001 Oct;51(4):740-6. doi: 10.1097/00005373-200110000-00020. PMID 11586169
- [Result] Hart DW, Wolf SE, Mlcak R, Chinkes DL, Ramzy PI, Obeng MK, Ferrando AA, Wolfe RR, Herndon DN. Persistence of muscle catabolism after severe burn. Surgery. 2000 Aug;128(2):312-9. doi: 10.1067/msy.2000.108059. PMID 10923010
- [Result] Ferrando AA, Lane HW, Stuart CA, Davis-Street J, Wolfe RR. Prolonged bed rest decreases skeletal muscle and whole body protein synthesis. Am J Physiol. 1996 Apr;270(4 Pt 1):E627-33. doi: 10.1152/ajpendo.1996.270.4.E627. PMID 8928769
- [Result] Ferrando AA, Paddon-Jones D, Wolfe RR. Bed rest and myopathies. Curr Opin Clin Nutr Metab Care. 2006 Jul;9(4):410-5. doi: 10.1097/01.mco.0000232901.59168.e9. PMID 16778570
- [Result] Bassey EJ, Bennett T, Birmingham AT, Fentem PH, Fitton D, Goldsmith R. Effects of surgical operation and bed rest on cardiovascular responses to exercise in hospital patients. Cardiovasc Res. 1973 Sep;7(5):588-92. doi: 10.1093/cvr/7.5.588. No abstract available. PMID 4753294
- [Result] Convertino V, Hung J, Goldwater D, DeBusk RF. Cardiovascular responses to exercise in middle-aged men after 10 days of bedrest. Circulation. 1982 Jan;65(1):134-40. doi: 10.1161/01.cir.65.1.134. PMID 6796287
- [Result] Convertino VA, Bisson R, Bates R, Goldwater D, Sandler H. Effects of antiorthostatic bedrest on the cardiorespiratory responses to exercise. Aviat Space Environ Med. 1981 Apr;52(4):251-5. No abstract available. PMID 7283897
- [Result] Greenleaf JE, Wade CE, Leftheriotis G. Orthostatic responses following 30-day bed rest deconditioning with isotonic and isokinetic exercise training. Aviat Space Environ Med. 1989 Jun;60(6):537-42. PMID 2751583
- [Result] Hung J, Goldwater D, Convertino VA, McKillop JH, Goris ML, DeBusk RF. Mechanisms for decreased exercise capacity after bed rest in normal middle-aged men. Am J Cardiol. 1983 Jan 15;51(2):344-8. doi: 10.1016/s0002-9149(83)80063-0. PMID 6823849
- [Result] Miller PB, Johnson RL, Lamb LE. Effects of moderate physical exercise during four weeks of bed rest on circulatory functions in man. Aerosp Med. 1965 Nov;36(11):1077-82. No abstract available. PMID 5860109
- [Result] Convertino V, Hoffler GW. Cardiovascular physiology. Effects of microgravity. J Fla Med Assoc. 1992 Aug;79(8):517-24. PMID 1402772
- [Result] Convertino VA. Effects of exercise and inactivity on intravascular volume and cardiovascular control mechanisms. Acta Astronaut. 1992 Jul;27:123-9. doi: 10.1016/0094-5765(92)90188-o. PMID 11537577
- [Result] Dudley GA, Gollnick PD, Convertino VA, Buchanan P. Changes of muscle function and size with bedrest. Physiologist. 1989 Feb;32(1 Suppl):S65-6. No abstract available. PMID 2727110
- [Result] Greenleaf JE, Van Beaumont W, Convertino VA, Starr JC. Handgrip and general muscular strength and endurance during prolonged bedrest with isometric and isotonic leg exercise training. Aviat Space Environ Med. 1983 Aug;54(8):696-700. No abstract available. PMID 6626077
- [Result] LeBlanc A, Gogia P, Schneider V, Krebs J, Schonfeld E, Evans H. Calf muscle area and strength changes after five weeks of horizontal bed rest. Am J Sports Med. 1988 Nov-Dec;16(6):624-9. doi: 10.1177/036354658801600612. PMID 3239619
- [Result] Bienso RS, Ringholm S, Kiilerich K, Aachmann-Andersen NJ, Krogh-Madsen R, Guerra B, Plomgaard P, van Hall G, Treebak JT, Saltin B, Lundby C, Calbet JA, Pilegaard H, Wojtaszewski JF. GLUT4 and glycogen synthase are key players in bed rest-induced insulin resistance. Diabetes. 2012 May;61(5):1090-9. doi: 10.2337/db11-0884. Epub 2012 Mar 8. PMID 22403297
- [Result] Stremel RW, Convertino VA, Bernauer EM, Greenleaf JE. Cardiorespiratory deconditioning with static and dynamic leg exercise during bed rest. J Appl Physiol. 1976 Dec;41(6):905-9. doi: 10.1152/jappl.1976.41.6.905. PMID 1002644
- [Result] Crandall CG, Shibasaki M, Wilson TE, Cui J, Levine BD. Prolonged head-down tilt exposure reduces maximal cutaneous vasodilator and sweating capacity in humans. J Appl Physiol (1985). 2003 Jun;94(6):2330-6. doi: 10.1152/japplphysiol.00790.2002. Epub 2003 Feb 21. PMID 12598483
- [Result] Greenleaf JE, Reese RD. Exercise thermoregulation after 14 days of bed rest. J Appl Physiol Respir Environ Exerc Physiol. 1980 Jan;48(1):72-8. doi: 10.1152/jappl.1980.48.1.72. PMID 7353981
- [Result] Levine DS, Greenleaf JE. Immunosuppression during spaceflight deconditioning. Aviat Space Environ Med. 1998 Feb;69(2):172-7. PMID 9491259
- [Result] Tipton CM, Greenleaf JE, Jackson CG. Neuroendocrine and immune system responses with spaceflights. Med Sci Sports Exerc. 1996 Aug;28(8):988-98. doi: 10.1097/00005768-199608000-00009. PMID 8871909
- [Result] DeRoshia CW, Greenleaf JE. Performance and mood-state parameters during 30-day 6 degrees head-down bed rest with exercise training. Aviat Space Environ Med. 1993 Jun;64(6):522-7. PMID 8338499
- [Result] Natelson BH, Deroshia C, Adamus J, Finnegan MB, Levin BE. Relations between visceral and behavioral function in men at bedrest. Pavlov J Biol Sci. 1983 Jul-Sep;18(3):161-8. doi: 10.1007/BF03019168. PMID 6622073
- [Result] Kress JP. Clinical trials of early mobilization of critically ill patients. Crit Care Med. 2009 Oct;37(10 Suppl):S442-7. doi: 10.1097/CCM.0b013e3181b6f9c0. PMID 20046133
- [Result] Stiller K. Physiotherapy in intensive care: an updated systematic review. Chest. 2013 Sep;144(3):825-847. doi: 10.1378/chest.12-2930. PMID 23722822
- [Result] Burnsworth B, Krob MJ, Langer-Schnepp M. Immediate ambulation of patients with lower-extremity grafts. J Burn Care Rehabil. 1992 Jan-Feb;13(1):89-92. PMID 1572864
- [Result] Grube BJ, Engrav LH, Heimbach DM. Early ambulation and discharge in 100 patients with burns of the foot treated by grafts. J Trauma. 1992 Nov;33(5):662-4. doi: 10.1097/00005373-199211000-00011. PMID 1361207
- [Result] General Principles of Exercise Prescription, in ACSM's Guidelines for Exercise Testing and Prescription, B.A. Franklin, Editor 2006, Lippincott Williams & Wilkins: Philadelphia.
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Result] Branski LK, Norbury WB, Herndon DN, Chinkes DL, Cochran A, Suman O, Benjamin D, Jeschke MG. Measurement of body composition in burned children: is there a gold standard? JPEN J Parenter Enteral Nutr. 2010 Jan-Feb;34(1):55-63. doi: 10.1177/0148607109336601. Epub 2009 Nov 2. PMID 19884353
- [Result] Herndon DN, Hart DW, Wolf SE, Chinkes DL, Wolfe RR. Reversal of catabolism by beta-blockade after severe burns. N Engl J Med. 2001 Oct 25;345(17):1223-9. doi: 10.1056/NEJMoa010342. PMID 11680441
- [Result] Przkora R, Herndon DN, Suman OE. The effects of oxandrolone and exercise on muscle mass and function in children with severe burns. Pediatrics. 2007 Jan;119(1):e109-16. doi: 10.1542/peds.2006-1548. Epub 2006 Nov 27. PMID 17130281
- [Result] Suman OE, Spies RJ, Celis MM, Mlcak RP, Herndon DN. Effects of a 12-wk resistance exercise program on skeletal muscle strength in children with burn injuries. J Appl Physiol (1985). 2001 Sep;91(3):1168-75. doi: 10.1152/jappl.2001.91.3.1168. PMID 11509512
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Brooks D, Solway S, Gibbons WJ. ATS statement on six-minute walk test. Am J Respir Crit Care Med. 2003 May 1;167(9):1287. doi: 10.1164/ajrccm.167.9.950. No abstract available. PMID 12714344
- [Result] Bartholomew K, Horowitz LM. Attachment styles among young adults: a test of a four-category model. J Pers Soc Psychol. 1991 Aug;61(2):226-44. doi: 10.1037//0022-3514.61.2.226. PMID 1920064
- [Result] Bartholomew, K. and E. Scharfe, Reliability and stability of adult attachment patterns. Personal relationships. J Pers Soc Psychol, 1994. 1: p. 23-43.